CLINICAL TRIAL: NCT06336096
Title: A Phase 1, Open-label, Randomized, Crossover Study to Evaluate the Relative Bioavailability and Food Effect of a New Tablet Formulation of Suzetrigine in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Relative Bioavailability and Food Effect of a New Tablet Formulation and Strength of Suzetrigine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VX23-548-017
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Participants will be randomized to receive a single dose of SUZ in 1 of 6 treatment sequences with 3 dosing periods to assess the relative bioavailability of two tablet formulations and the effect of food on the PK of SUZ. There will be a 14-day washout period between each dosing period.
  Interventions: Drug: Suzetrigine
- Part B (Experimental): Participants will be randomized to receive a single dose of SUZ formulation in 1 of 2 treatment sequences with 2 dosing periods to assess the relative bioavailability of tablet formulation compared to a suspension of SUZ. There will be a 14-day washout period between each dosing period.
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Tablet(s) for oral administration.
  Other Names: VX-548; SUZ
  Arms: Part A
Drug: Suzetrigine — Tablet(s) and Suspension for oral administration.
  Other Names: VX-548; SUZ
  Arms: Part B

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of suzetrigine (SUZ; VX-548) and its metabolite along with its safety and tolerability, in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (Kg/m^2)
* A total body weight greater than (>) 50 kilogram (kg)
* Participants of non-childbearing potential

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of SUZ | Pre-dose up to Day 43
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-tlast) of SUZ | Pre-dose up to Day 43
Part A: Area Under the Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of SUZ | Pre-dose up to Day 43
Part B: Cmax of SUZ | Pre-dose up to Day 29
Part B: AUC0-tlast of SUZ | Pre-dose up to Day 29
Part B: AUC0-inf of SUZ | Pre-dose up to Day 29

SECONDARY OUTCOMES:
Part A: Cmax of SUZ Metabolite | Pre-dose up to Day 43
Part A: AUC0-tlast of SUZ Metabolite | Pre-dose up to Day 43
Part A: AUC0-inf of SUZ Metabolite | Pre-dose up to Day 43
Part A: Safety and Tolerability as Assessed by Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 43
Part B: Cmax of SUZ Metabolite | Pre-dose up to Day 29
Part B: AUC0-tlast of SUZ Metabolite | Pre-dose up to Day 29
Part B: AUC0-inf of SUZ Metabolite | Pre-dose up to Day 29
Part B: Safety and Tolerability as Assessed by Number of Participants with AEs and SAEs | From Day 1 up to Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion - Tempe, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing